CLINICAL TRIAL: NCT02576639
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Oral Doses of CNP520 in Healthy Elderly Subjects
Brief Title: Dose-ranging Safety and Tolerability Study in Subjects ≥60 Years of Age
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: CCNP520X2102; 2013-005576-18 (EudraCT Number)
Record Dates: First submitted 2015-08-18; First posted 2015-10-15 (Estimated); Results first posted 2017-05-25 (Actual); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease,; Amyloid Beta,; cerebrospinal fluid,; beta secretase
MeSH Terms: conditions — Alzheimer Disease; Plaque, Amyloid | interventions — Umibecestat; Capsules

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (5):
- Placebo (Placebo Comparator): Matching placebo to CNP520 was taken once daily (qd) orally for 13 weeks.
  Interventions: Drug: Placebo
- CNP520 2 mg (Experimental): CNP520 2 mg was taken qd orally for 13 weeks.
  Interventions: Drug: CNP520
- CNP520 10 mg (Experimental): CNP520 10 mg was taken qd orally for 13 weeks.
  Interventions: Drug: CNP520
- CNP520 35 mg (Experimental): CNP520 35 mg was taken qd orally for 13 weeks.
  Interventions: Drug: CNP520
- CNP520 85 mg (Experimental): CNP520 85 mg was taken qd orally for 13 weeks.
  Interventions: Drug: CNP520

INTERVENTIONS:
Drug: CNP520
  Other Names: CNP520 was supplied as capsules in dose strengths of 1 mg, 10 mg, 25 mg and 75 mg.
  Arms: CNP520 10 mg; CNP520 2 mg; CNP520 35 mg; CNP520 85 mg
Drug: Placebo — Matching placebo to CNP520 was supplied in capsules.
  Arms: Placebo

SUMMARY:
The study determined the safety of CNP520 in healthy elderly over 3 months. Data relevant for Pharmacokinetic/Pharmacodynamic modeling were obtained in order to define the target dose in subsequent efficacy studies.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy status
* Body weight: ≥45kg
* BMI: 18-34 kg/m2

Key Exclusion Criteria:

* History or presence of any clinically significant disease of any major system organ class.
* Heavy smoker status
* History /presence of clinically significant neurological or psychiatric disorders
* Any medical condition that might lead to or is associated with any cognitive deficit
* History or presence of severely impaired renal function

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2015-08-10 (Actual); Primary Completion 2016-03-11 (Actual); Study Completion 2016-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Novartis Pharmaceuticals
Locations (11):
- United States (4):
  - Novartis Investigative Site, Glendale, California
  - Novartis Investigative Site, Long Beach, California
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Lincoln, Nebraska
- Novartis Investigative Site, Antwerp, Belgium
- Novartis Investigative Site, Berlin, Germany
- Netherlands (2):
  - Novartis Investigative Site, Groningen, GZ
  - Novartis Investigative Site, Leiden
- United Kingdom (3):
  - Novartis Investigative Site, Belfast, Northern Ireland
  - Novartis Investigative Site, Harrow
  - Novartis Investigative Site, Mid Glamorgan

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized in a 1:1:1:1:1 ratio to 5 treatment groups: placebo, CNP520 2 mg, CNP520 10 mg, CNP520 35 mg and CNP520 85 mg.
Period: Overall Study
Arm/Group | Placebo | CNP520 2 mg | CNP520 10 mg | CNP520 35 mg | CNP520 85 mg
Started | 24 | 25 | 25 | 26 | 24
Pharmacodynamic Analysis Set | 24 | 24 | 25 | 25 | 25
Pharmacokinetic Analysis Set | 0 | 25 | 25 | 26 | 24
Safety Analysis Set | 24 | 25 | 25 | 26 | 24
Completed | 22 | 23 | 23 | 25 | 20
Not Completed | 2 | 2 | 2 | 1 | 4
Not completed — Withdrawal by Subject | 1 | 2 | 1 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 1 | 1 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | CNP520 2 mg | CNP520 10 mg | CNP520 35 mg | CNP520 85 mg | Total
Number analyzed (Participants) | 24 | 25 | 25 | 26 | 24 | 124
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.6 (5.3) | 65.4 (4.6) | 66.8 (5.1) | 66.1 (4.6) | 66.5 (5.2) | 66.3 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 16 | 13 | 11 | 9 | 61
  Male | 12 | 9 | 12 | 15 | 15 | 63

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Non-serious and Serious Adverse Events (AEs) and Deaths
Description: Safety monitoring was conducted throughout the study.
Time Frame: 13 weeks
Population: The safety analysis set, which included participants who received at least 1 dose of study drug (CNP520 or placebo), was analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | CNP520 2 mg | CNP520 10 mg | CNP520 35 mg | CNP520 85 mg
Number analyzed (Participants) | 24 | 25 | 25 | 26 | 24
Participants
  Non-serious AEs | 18 | 19 | 22 | 20 | 18
  Serious AEs | 0 | 0 | 0 | 1 | 0
  Deaths | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Change From Baseline of Amyloid Beta (Aβ) 1-38 , Aβ 1-40 and Aβ 1-42 Cerebrospinal Fluid (CSF) Concentrations
Description: CSF samples were collected by lumbar puncture for assessment.
Time Frame: Day 92
Population: The pharmacodynamics (PD) analysis set was analyzed. The PD set included only randomized participants who had available PD data and no protocol deviations with relevant impact on PD data.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Placebo | CNP520 2 mg | CNP520 10 mg | CNP520 35 mg | CNP520 85 mg
Number analyzed (Participants) | 21 | 22 | 21 | 23 | 20
Percentage change
  Aβ 1-38 | -2.34 (6.969) | -20.55 (10.475) | -62.48 (6.202) | -82.93 (4.378) | -89.5 (1.676)
  Aβ 1-40 | -2.64 (6.598) | -22.64 (9.937) | -62.89 (6.485) | -83.16 (4.227) | -90.69 (1.651)
  Aβ 1-42 | -2.58 (5.189) | -23.93 (8.987) | -64.28 (6.086) | -82.35 (5.474) | -89.68 (2.32)

3. Secondary Outcome: Summary of Plasma PK Parameter: Cmax
Description: Cmax = the observed maximum plasma concentration following drug administration. Blood samples were collected to assess Cmax. The PK analysis set was used for the analysis.
Time Frame: Days 1, 91
Population: The PK analysis set was used for the analysis. For a given time point, only those participants from the PK analysis set, who had PK data and had no protocol deviations with relevant impact on PK data, were analyzed for that time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CNP520 2 mg | CNP520 10 mg | CNP520 35 mg | CNP520 85 mg
Number analyzed (Participants) | 25 | 25 | 26 | 24
ng/mL
  Day 1 (n=25,25,26,24) | 4.76 (2.92) | 21.3 (6.67) | 75.6 (23.4) | 163 (47.4)
  Day 91 (=23,22,24,20) | 16.6 (5.51) | 81 (29.2) | 237 (65.7) | 602 (150)

4. Secondary Outcome: Summary of Plasma PK Parameter: AUCtau
Description: AUCtau = the area under the plasma concentration-time curve from zero to the end of the dosing interval tau. Blood samples were collected to assess AUCtau.
Time Frame: Days 1 and 91
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | CNP520 2 mg | CNP520 10 mg | CNP520 35 mg | CNP520 85 mg
Number analyzed (Participants) | 25 | 25 | 26 | 24
h*ng/mL
  Day 1 (n=25,25,26,24) | 67.1 (60.7) | 278 (65.7) | 966 (214) | 2300 (479)
  Day 91 (n=23,22,24,20) | 313 (117) | 1500 (476) | 4450 (1090) | 11200 (3320)

5. Secondary Outcome: Summary of Plasma PK Parameter: Tmax
Description: Tmax = the time to reach the maximum concentration after drug administration. Blood samples were collected to assess Tmax.
Time Frame: Days 1 and 91
Population: as for outcome 3
Measure: Median (Full Range); unit: hour
Arm/Group | CNP520 2 mg | CNP520 10 mg | CNP520 35 mg | CNP520 85 mg
Number analyzed (Participants) | 25 | 25 | 26 | 24
hour
  Day 1 (n=25,25,26,24) | 2.5 [2.45 to 9] | 2.5 [2.5 to 6.02] | 2.5 [2.48 to 9] | 2.5 [2.42 to 12]
  Day 91 (n=23,22,24,20) | 2.5 [0 to 12.1] | 2.5 [0 to 12.5] | 2.5 [0 to 12] | 2.5 [0 to 12]

6. Secondary Outcome: Summary of Plasma PK Parameter: Tlag
Description: Tlag = time delay between drug administration and first observed concentration above the lower limit of quantification (LOQ) in plasma . Blood samples were collected to assess Tlag.
Time Frame: Days 1 and 91
Population: as for outcome 3
Measure: Median (Full Range); unit: hour
Arm/Group | CNP520 2 mg | CNP520 10 mg | CNP520 35 mg | CNP520 85 mg
Number analyzed (Participants) | 25 | 25 | 26 | 24
hour
  Day 1 (n=25,25,26,24) | 0.5 [0 to 0.567] | 0.5 [0 to 2.5] | 0.5 [0 to 0.55] | 0 [0 to 2.5]
  Day 91 (n=23,22,24,20) | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

7. Secondary Outcome: Summary of Plasma PK Parameter: T1/2
Description: T1/2 = the terminal elimination half-life. Blood samples were collected to assess T/12.
Time Frame: Day 91
Population: The PK analysis set was used for the analysis. Only those participants from the PK analysis set, who had PK data and had no protocol deviations with relevant impact on PK data, were analyzed.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | CNP520 2 mg | CNP520 10 mg | CNP520 35 mg | CNP520 85 mg
Number analyzed (Participants) | 23 | 22 | 24 | 20
hour | 150 (52.2) | 155 (40.9) | 155 (33.9) | 160 (22)

8. Secondary Outcome: Summary of PK Parameter: CLss/F
Description: CLss/F = the apparent systemic clearance from plasma observed during a dosing interval at steady state following extravascular administration. Blood samples were collected to assess CLss/F.
Time Frame: Day 91
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mL/h
Arm/Group | CNP520 2 mg | CNP520 10 mg | CNP520 35 mg | CNP520 85 mg
Number analyzed (Participants) | 23 | 22 | 24 | 20
mL/h | 7620 (2620) | 7380 (2480) | 8460 (2790) | 8220 (2270)

9. Secondary Outcome: Summary of Plasma PK Parameter: Racc
Description: Racc = the accumulation ratio . Blood samples were collected to assess Racc.
Time Frame: Day 91
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | CNP520 2 mg | CNP520 10 mg | CNP520 35 mg | CNP520 85 mg
Number analyzed (Participants) | 23 | 22 | 24 | 20
ratio | 5.86 (2.25) | 5.33 (1.05) | 4.75 (1.16) | 5.02 (1.47)

10. Secondary Outcome: Summary of CSF PK Concentrations
Description: CSF samples were collected by lumbar puncture for assessment.
Time Frame: Days 1, 14, 28, 42, 56, 70 and 91
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CNP520 2 mg | CNP520 10 mg | CNP520 35 mg | CNP520 85 mg
Number analyzed (Participants) | 25 | 25 | 26 | 24
ng/mL
  Day 1 (n=24,25,26,24) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Day 14 (n=3,4,4,4) | 0.166 (0.103) | 1.07 (0.225) | 3.82 (0.868) | 8.13 (2.7)
  Day 28 (n=5,2,7,5) | 0.303 (0.0731) | 1.48 (0.106) | 4.48 (1.02) | 12 (4.12)
  Day 42 (n=3,6,5,5) | 0.314 (0.0715) | 1.52 (0.6) | 4 (1.21) | 7.47 (1.57)
  Day 56 (n=5,5,2,4) | 0.291 (0.0605) | 1.28 (0.177) | 5.03 (2.69) | 8.04 (5.69)
  Day 70 (n=6,5,6,4) | 0.231 (0.149) | 1.04 (0.212) | 4.62 (0.753) | 8.71 (0.71)
  Day 91 (n=23,21,24,20) | 0.305 (0.099) | 1.44 (0.431) | 4.52 (0.946) | 10.4 (3.26)

11. Secondary Outcome: Area-under-plasma Concentration Time Curve up to Infinity (AUCinf)
Description: CNP520 concentrations in plasma
Time Frame: Day 91
Population: This PK parameter was not analyzed because data was not collected.
Arm/Group | CNP520 2 mg | CNP520 10 mg | CNP520 35 mg | CNP520 85 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

12. Secondary Outcome: Apparent Volume of Distribution (Vz/F)
Time Frame: Day 91
Population: This PK parameter was not analyzed because data was not collected.
Arm/Group | CNP520 2 mg | CNP520 10 mg | CNP520 35 mg | CNP520 85 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Groups:
- CNP520 2mg: CNP520 2 mg was taken qd orally for 13 weeks.
- CNP520 10mg: CNP520 10 mg was taken qd orally for 13 weeks.
- CNP520 35mg: CNP520 35 mg was taken qd orally for 13 weeks.
- CNP520 85mg: CNP520 85 mg was taken qd orally for 13 weeks.
Arm/Group | Placebo | CNP520 2mg | CNP520 10mg | CNP520 35mg | CNP520 85mg
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/25 | 0/25 | 1/26 | 0/24
Other Adverse Events (participants affected / at risk) | 18/24 | 19/25 | 22/25 | 20/26 | 18/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=24) | CNP520 2mg (N=25) | CNP520 10mg (N=25) | CNP520 35mg (N=26) | CNP520 85mg (N=24)
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=24) | CNP520 2mg (N=25) | CNP520 10mg (N=25) | CNP520 35mg (N=26) | CNP520 85mg (N=24)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 1 | 0
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Asthenopia (Eye disorders) | 0 | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 1
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 1
Eye pain (Eye disorders) | 0 | 0 | 1 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 2 | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 0 | 1 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 1 | 0 | 0 | 1
Vision blurred (Eye disorders) | 1 | 1 | 2 | 0 | 1
Visual impairment (Eye disorders) | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 5 | 1 | 3 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 2 | 1 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Faeces hard (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Faeces soft (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 1 | 3 | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 3 | 2 | 2
Toothache (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2 | 0 | 2 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 3 | 0 | 0 | 2 | 2
Feeling cold (General disorders) | 0 | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 1
Injection site pain (General disorders) | 0 | 0 | 0 | 1 | 2
Pain (General disorders) | 0 | 0 | 1 | 0 | 0
Puncture site pain (General disorders) | 0 | 1 | 1 | 1 | 0
Vessel puncture site haemorrhage (General disorders) | 1 | 0 | 1 | 0 | 0
Vessel puncture site pain (General disorders) | 0 | 0 | 1 | 0 | 0
Vessel puncture site swelling (General disorders) | 0 | 0 | 1 | 0 | 0
Allergy to chemicals (Immune system disorders) | 0 | 0 | 0 | 0 | 1
Abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Abscess jaw (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Hordeolum (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 4 | 2 | 5 | 4 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Tinea pedis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 2 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Ear abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Foreign body in eye (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 2 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 8 | 2 | 1 | 3 | 3
Post procedural discomfort (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 1
Procedural dizziness (Injury, poisoning and procedural complications) | 2 | 0 | 3 | 2 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 3 | 4 | 2 | 3
Scratch (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Traumatic lumbar puncture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Amylase increased (Investigations) | 0 | 1 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 2 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 1 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3 | 3 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 2 | 2 | 3 | 4
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 1 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 2 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 1 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 1 | 1 | 0 | 1
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 0 | 1 | 1 | 0
Dizziness postural (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Head discomfort (Nervous system disorders) | 1 | 1 | 1 | 0 | 0
Headache (Nervous system disorders) | 10 | 11 | 5 | 5 | 5
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Sedation (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 1 | 0 | 2 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Visual field defect (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 1 | 1 | 1 | 1
Affective disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Irritability (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Libido decreased (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Nightmare (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Obsessive thoughts (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 1
Polyuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Pruritus genital (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3 | 3 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 2 | 2 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 1 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 0 | 1 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.